CLINICAL TRIAL: NCT05476250
Title: Clinical Performance of Masimo INVSENSOR00057 for Atrial Fibrillation Detection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The validation protocol is no longer needed for regulatory submission.
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1022
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00057 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00057.
  Interventions: Device: INVSENSOR00057

INTERVENTIONS:
Device: INVSENSOR00057 — Noninvasive wearable health monitoring device

SUMMARY:
This study is designed to validate the performance of Masimo INVSENSOR00057 in detecting atrial fibrillation. The noninvasive ECG measurements will be compared to results obtained from an FDA-cleared ECG monitor.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 to 80 years of age.
* Subject can read and communicate in English.
* Subject's cardiac rhythm shall be Normal Sinus Rhythm or Atrial Fibrillation (Afib). This determination will be made using FDA cleared 3-lead ECG which will label subject's cardiac rhythm as such.

Exclusion Criteria:

* Subject has open wounds, inflamed tattoos or piercings on the area of device placement, and/or has any visible healing wounds that the investigator and/or medical professional determines may place them at an increased risk for participation.
* Subject has any medical condition which in the judgment of the investigator and/or study staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Masimo INVSENSOR00057: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00057.
  INVSENSOR00057: Noninvasive wearable health monitoring device
Period: Overall Study
Arm/Group | Masimo INVSENSOR00057
Started | 120
Completed | 99
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Masimo INVSENSOR00057
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 34
  More than one race | 7
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Specificity of Masimo INVSENSOR00057 Atrial Fibrillation Detection Function
Description: Specificity refers to the ability of Masimo INVSENSOR00057 to correctly identify individuals who do not have atrial fibrillation. High specificity is important in minimizing false positives.
Time Frame: 1-5 hours
Population: 1 subject not analyzed due to EDC error.
Measure: Number; unit: % of true negatives
Arm/Group | Masimo INVSENSOR00057
Number analyzed (Participants) | 98
% of true negatives | 100

ADVERSE EVENTS:
Time Frame: 1-5 hours
Arm/Group | Masimo INVSENSOR00057
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT05476250/Prot_SAP_000.pdf